CLINICAL TRIAL: NCT02586428
Title: Decision-Making in Patients Regarding Noninvasive Prenatal Testing
Brief Title: Noninvasive Prenatal Testing
Status: Terminated | Type: Observational
Why Stopped: difficult to enroll, Pi decision to closed
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, fruhman@slu.edu, PI, St. Louis University
Other Study IDs: 25878
Record Dates: First submitted 2015-09-08; First posted 2015-10-26 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Genetic Counseling

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: what patients elect noninvasive prenatal testing (NIPT) — what percentages of patients elect noninvasive prenatal testing (NIPT), amniocentesis, or no testing before and after genetic counseling.

SUMMARY:
Before and after a patient receives genetic counseling they will be offered the chance to complete the survey, by their counselor. Since each patient sees only one genetic counselor that counselor will be responsible for consenting and giving and collecting the finish surveys. No identifiers will be used. The investigators will emphasize that their answers will remain anonymous throughout the entire process, and that their participation is strictly voluntary. The patient will be provided with a survey and asked to complete this before their genetic counseling session and after.The survey will be returned to the genetic counselor and placed in a locked drawer. Information will also be collected from the medical record including age, pregnancy history and the reason for the visit.

DETAILED DESCRIPTION:
Patients who have abnormal ultrasound findings,advanced maternal age, abnormal serum biochemical screening, or a personal or family history of chromosomal/genetic conditions will be eligible for this study. Prior to receiving genetic counseling, the genetic counselor or her designee will approach the patient asking if she would be willing to participate in a survey that helps us better determine how well patients understand their testing options for the above issues.

The survey consists of two parts. The first part will be taken prior to genetic counseling to see what the patient's baseline understanding of their options are (this is study related.) If the patient agrees to participate in the study, she will then receive the first part of the survey. After completion of the first part of the survey, the patient will then receive genetic counseling (this is standard of care.). Information will also be collected from the medical record including age, pregnancy history and the reason for the visit. After receiving genetic counseling for their specific indication, patients will decide if they want noninvasive prenatal testing, amniocentesis, testing depending what their ultrasound shows, or no testing. After this the patient will be given the second part of the survey to complete (this is study related). Regardless of which testing is elected, (if any), participants are administered the same survey. After completing the survey, the patient will return the form to the genetic counselor or her designee. The recruitment period is expected to last approximately one year. After recruitment is completed, data analysis will take place. Interim data analysis make take place as well.

Patients will not be contacted for research purposes after the survey has been completed.

After patients complete this survey, they will require no further information. They are not being administered a treatment or receiving a direct benefit from participation; the study is designed only to obtain information about patient's decisions, knowledge, and attitudes regarding their testing options.

ELIGIBILITY:
Inclusion Criteria:

* high risk pregnant women seen for genetic counseling

Exclusion Criteria:

* low risk
* not pregnant

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have abnormal ultrasound findings, advance maternal age, abnormal serum biochemical screening, or a personal or family history of chromosomal/genetic conditions will be eligible for this study. These patients will be scheduled ahead of time with the genetic counseling.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
will measure what percentages of patients elect noninvasive prenatal testing (NIPT), amniocentesis, or no testing before and after genetic counseling | over the next 6 months
  percentages of patient's choices

SECONDARY OUTCOMES:
will measure patients' reasons for electing or not electing testing | over the next 6 months
  Reasons for not electing to have testing
Measure if patients' understand the different testing options. | over next 6 months
  Are they able to give explanation of testing

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fruhman, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Hospital, St Louis, Missouri, United States